CLINICAL TRIAL: NCT03892018
Title: An Open-label, Crossover Study of the Effect of Food on the Pharmacokinetics of Paclitaxel Administered Orally as Oraxol
Brief Title: The Effect of Food on the Pharmacokinetics of Paclitaxel Administered Orally as Oraxol
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: STUDY HALTED DUE TO FINANCIAL CONTRAINTS
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-012
Record Dates: First submitted 2019-03-19; First posted 2019-03-27 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: This will be an open-label, 2-part, crossover study to assess the effect of food on Oraxol exposure. The study will consist of the following periods: Screening, Baseline, Periods 1 and 2 (Part A), Treatment (Part B), and Follow-up. Part A will assess the effect of food on Oraxol pharmacokinetics. In Part A, subjects will be randomized to the sequence (fed/fasted or fasted/fed conditions) under which they will be administered single-dose treatment after an overnight fast. There will be a minimum of 7 days after Period 1 treatment before subjects cross over to Period 2 treatment. Subjects who have participated in the PK assessments in Part A of the study may continue into Part B, during which Oraxol will be dosed for 3 consecutive days per week under fasting conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fed/ Fasted Treatment Sequence (Active Comparator): Subjects will be assigned a fed/fasted sequence.
  Fed sequence- subjects will fast overnight and continue fasting until they consume a standardized test meal at a predetermined time after paclitaxel administration.
  Fasted Sequence- subjects will fast overnight and continue fasting until 4 hours post paclitaxel dose.
  Interventions: Drug: Oraxol
- Fasted/ Fed Treatment Sequence (Active Comparator): Subjects will be assigned a fasted/fed sequence.
  Fasted Sequence- subjects will fast overnight and continue fasting until 4 hours post paclitaxel dose.
  Fed sequence- subjects will fast overnight and continue fasting until they consume a standardized test meal at a predetermined time after paclitaxel administration.
  Interventions: Drug: Oraxol

INTERVENTIONS:
Drug: Oraxol — Oraxol will be supplied as paclitaxel capsules and HM30181AK-US tablets.
  Other Names: Paclitaxel and HM30181AK-US

SUMMARY:
This is multicenter, open-label, 2-part crossover study. Eligible subjects will have metastatic or unresectable solid tumors. This study includes a pretreatment and treatment phase. The pretreatment phase consists of screening and baseline. The treatment phase consists of Periods 1 and 2 (Part A), Treatment (Part B), and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Measurable disease as per RECIST v1.1 criteria
* Adequate hematologic status
* Adequate liver function.
* Adequate renal function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy of at least 3 months.
* Women must be postmenopausal or surgically sterile.
* Sexually active male subjects must use a barrier method of contraception during the study.
* Able to consume the prescribed meals

Exclusion Criteria:

* Have not recovered to ≤ Grade 1 toxicity from previous anticancer treatments or previous investigational products (IPs).
* Received IPs within 21 days or 5 half-lives of the first dosing day, whichever is shorter
* Are currently receiving other medications or radiation intended for the treatment of their malignancy. Hormonal therapy is allowed.
* Women of childbearing potential who are pregnant or breastfeeding.
* Currently taking a concomitant medication, other than a premedication, that is:

  * A strong P-glycoprotein (P-gp) inhibitor or inducer.
  * An oral medication with a narrow therapeutic index known to be a P-gp substrate.
  * Medications known to be strong inhibitors or inducers of cytochrome P450 (CYP) 2C8 or medications known to be strong CYP3A4 inhibitors or inducers.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or any concomitant illness that would limit compliance with study requirements.
* Major surgery to the upper gastrointestinal (GI) tract, or have a history of GI disease that may interfere with oral drug absorption.
* Cirrhosis of the liver or known active hepatitis B, hepatitis C, or HIV
* History of hypersensitivity to paclitaxel, not attributed to a hypersensitivity-type reaction to Cremophor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the concentration-time profile of Oral Paclitaxel in plasma for 168 hours when taken with or without food. | 24 months

SECONDARY OUTCOMES:
Comparison of the concentration-time profile of HM30181 in plasma for 168 hours when taken with or without food. | 24 months
The proportion of patients with tumor responses after the initiation of treatment. | At baseline and every 8 weeks through study completion, approximately 24 months
  RECIST v1.1 criteria defined as complete response, partial response, stable disease or progressive disease
Incidence of Adverse Events (Safety and Tolerability) | 24 months
  Evaluate the safety of Oraxol. Number of participants with treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Athenex, Inc.
Locations (3):
- United Kingdom (3):
  - The Beatson West of Scotland Cancer Care Centre, Glasgow
  - The Christie NHS Foundation Trust, Manchester
  - The Northern Institute for Cancer Care, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No